CLINICAL TRIAL: NCT05304598
Title: Randomized Case Control Study Using Dexmedetomidine Prior to Intubation in Neonates
Brief Title: Using Dexmedetomidine Prior to Intubation in Neonates
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not able to recruit patients due to lack of consent.
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Alok Bhutada, Principal Investigator, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-03-05
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Effect Neonatal
Keywords: sedation; intubation; neonates; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Group (Active Comparator): a single intravenous (i.v.) dose of dexmedetomidine, 0.2 mcg/kg over 10 minutes
  Interventions: Drug: Dexmedetomidine
- Control Group (Active Comparator): routine awake intubation as per current unit standard of care
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Dexmedetomidine — a single intravenous (i.v.) dose of dexmedetomidine, 0.2 mcg/kg over 10 minutes
  Arms: Dexmedetomidine Group
Other: Usual Care — routine awake intubation as per current unit standard of care,
  Arms: Control Group

SUMMARY:
Neonatal intubations are performed routinely in a NICU. Most intubations are still performed without the administration of medications (awake intubations). Some of the reasons are unavailability of a single good medication, the ease of administration, the physicians comfort level, side effects of medications including apnea, bradycardia, hypotension. Some units use a cocktail of different medications, each with their own side effects We are proposing to study the effects of a single medication, dexmedetomidine (precedex) for the purpose of sedation prior to intubation in neonates.

This study will compare the efficacy of a single dose of dexmedetomidine to controls.

DETAILED DESCRIPTION:
This is an interventional un-blinded, randomized, prospective pilot study to examine the efficacy of dexmedetomidine in reducing time to intubation, pain/discomfort associated with intubation and maintaining better oxygen saturations in neonates during intubation. The study will be done in the Neonatal Intensive Care Unit at Maimonides Medical Center.

Parents of babies requiring intubation will be approached by the Neonatal attending / fellow to obtain consent for the study. If a consent is obtained, babies will be randomized to a control or study group. Babies in the control group will undergo routine intubation by a neonatologist but with monitoring of the vital signs, those in the study group will receive the study drug 10 minutes prior to intubation.

Data Collection Procedures:

The research data will reside in an encrypted laptop issued by MIS that is housed in the Division of Newborn Medicine, within the medical center.

The data will be accessible to all researchers. If needed, de-identified data will be stored/shared on the Maimonides share point website for statistical and backup purposes.

The data that will be collected are heart rate, respiratory rate, oxygen saturation, measured continuously, and blood pressure measurement every five minutes. Data will be collected 15 minutes before, during and 30 minutes after intubation.

ELIGIBILITY:
Inclusion Criteria:

* neonates
* elective intubation
* admitted to the NICU
* Less than 44 weeks corrected gestational age requiring intubation

Exclusion Criteria:

* babies requiring emergent intubation
* Neonates with birth weight<1250 grams and <1 week of postnatal age
* Neonates with major congenital malformations
* Neonates with preexisting hypotension (MAP < Gest Age)
* Neonates with complex congenital heart disease and heart block

Ages: 0 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation Differences | 30 minutes
  Compare oxygen saturation differences between the control and study group

CONTACTS AND LOCATIONS:
Overall Officials: Alok Bhutada, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT05304598/Prot_SAP_000.pdf